CLINICAL TRIAL: NCT03019172
Title: Safety, and Effectiveness of Lactobacillus Reuteri for the Treatment of Urinary Tract Infections in Women: A Pilot Randomized Clinical Trial (RCT)
Brief Title: Clinical Trial of L. Reuteri in Urinary Tract Infections in Non Pregnant Women
Acronym: UTIReuteri
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovacion y Desarrollo de Estrategias en Salud (Other)
Responsible Party: Principal Investigator, Pedro Gutierrez Castrellon, MD, MSc, DSc, Innovacion y Desarrollo de Estrategias en Salud
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UTIReuteri2016
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, double blind allocation concealment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactobacillus reuteri (Experimental): Women in experimental branch will receive two sachets. Sachet one contains a total of 5*10^8 CFU of Lactobacillus reuteri DSM 16666 & Lactobacillus reuteri DSM 17938, mixed with maltodextrin for flowability during production. Sachet two contains instant cranberry drink composed of Cranberry extract, xylitol, cranberry aroma, monosodium citrate, zink gluconate, silica.
  Interventions: Combination Product: Lactobacillus reuteri
- Sachet with cranberry + placebo (Placebo Comparator): Women in control branch will receive two sachets. Sachet one contains only Maltodextrin and sachet two contains instant cranberry drinkcomposed of Cranberry extract, xylitol, cranberry aroma, monosodium citrate, zink gluconate, silica Both sachets should be emptied in a glass and mixed with 200 ml of cold water
  Interventions: Dietary Supplement: Sachet with cranberry + placebo

INTERVENTIONS:
Combination Product: Lactobacillus reuteri — Sachet one contains a total of 5*10^8 CFU of Lactobacillus reuteri DSM 16666 & Lactobacillus reuteri DSM 17938, mixed with maltodextrin for flowability during production. Sachet two contains instant cranberry drink composed of Cranberry extract, xylitol, cranberry aroma, monosodium citrate, zink gluconate, silica. The products will be taken twice per day, morning and evening. The daily dose in the active group will be at least 5*10^8 CFU of L.reuteri DSM16666 and L. reuteri DSM17938), PAC-A and zinc
  Arms: Lactobacillus reuteri
Dietary Supplement: Sachet with cranberry + placebo — Sachet one contains placebo for probiotics (maltodextrin). Sachet two contains instant cranberry drink composed of Cranberry extract, xylitol, cranberry aroma, monosodium citrate, zink gluconate, silica.
  Arms: Sachet with cranberry + placebo

SUMMARY:
RCT to evaluate the safety and efficacy of Lactobacillus reuteri DSM 16666 & Lactobacillus reuteri DSM 17938 to significantly modify the frequency of clinical or bacteriological cure in women with non complicated acute cystitis who receive probiotics for 12 days compared with the frequency in women who receive placebo.

DETAILED DESCRIPTION:
Randomized, double blind, placebo controlled, pilot trial to evaluate the safety and efficacy of L. reuteri in non menopausal women with non complicated cystitis in terms of the frequency of clinical or bacteriological cure. Secondary outcomes will be a) time to clinical/laboratory relapse in at least 70% of women with non complicated acute cystitis who receive probiotics for 12 days compared with the time in women who receive placebo; b) frequency of clinical/laboratory and bacteriologic relapse in women with non complicated acute cystitis who receive probiotics for 12 days compared with the frequency in women who receive placebo, at day 30 after treatment start and c) frequency of adverse related events in women with non complicated acute cystitis who receive probiotics for 12 days compared with the frequency in women who receive placebo. In the active product we will use 5*10^8 CFU of Lactobacillus reuteri DSM 16666 & Lactobacillus reuteri DSM 17938 + cranberry extract. The control group will recibe Cranberry extract. The products will be taken twice per day, morning and evening.

ELIGIBILITY:
Inclusion Criteria:

* Non pregnant pre menopausal women
* Minimum age 18 years
* Uncomplicated cystitis diagnosed by urine dipstick testing (nitrates +, leukocytes esterase

  * and/or 105 CFU/ml or nitrates +, leukocytes esterase + and/or 102 -103 CFU/ml+ clinical symptoms) and an evaluation of the presence of typical related symptoms. In particular, frequency (frequent voiding of urine), urgency (the urge to void immediately), dysuria (painful voiding), and/or suprapubic pain.
* Verbal and Written Informed Consent for participation in the study

Exclusion Criteria:

* Acute cystitis symptoms for >1week before the first visit
* Diabetes mellitus,
* Congenital urinary tract abnormality
* Lactating women
* Female who intend to become pregnant during the study or within 3 months after the completion of the study
* Vaginal discharge + fever (>37.5oC)
* Diagnostic of sexually transmitted diseases
* Use of an indwelling catheter or an intermittent self-catheterisation program
* Presence of neurogenic bladder, or
* Use of any antibiotic 2 weeks before Day 1 in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-03-05 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
clinical and bacteriological cure | 30 days
  Frequency of clinical or bacteriological cure in women with non complicated acute cystitis who receive probiotics for 12 days compared with the frequency in women who receive placebo

SECONDARY OUTCOMES:
clinical or bacteriological relapse | 30 days
  Time to clinical/laboratory relapse in at least 70% of women with non complicated acute cystitis who receive probiotics for 12 days compared with the time in women who receive placebo
Adverse events | 14 days
  • Frequency of adverse related events in women with non complicated acute cystitis who receive probiotics for 12 days compared with the frequency in women who receive placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Dr. Manuel Gea Gonzalez, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee BB, Toh SL, Ryan S, Simpson JM, Clezy K, Bossa L, Rice SA, Marial O, Weber G, Kaur J, Boswell-Ruys C, Goodall S, Middleton J, Tudehope M, Kotsiou G. Probiotics [LGG-BB12 or RC14-GR1] versus placebo as prophylaxis for urinary tract infection in persons with spinal cord injury [ProSCIUTTU]: a study protocol for a randomised controlled trial. BMC Urol. 2016 Apr 16;16:18. doi: 10.1186/s12894-016-0136-8. PMID 27084704
- [Background] Schwenger EM, Tejani AM, Loewen PS. Probiotics for preventing urinary tract infections in adults and children. Cochrane Database Syst Rev. 2015 Dec 23;2015(12):CD008772. doi: 10.1002/14651858.CD008772.pub2. PMID 26695595
- [Background] Chisholm AH. Probiotics in Preventing Recurrent Urinary Tract Infections in Women: A Literature Review. Urol Nurs. 2015 Jan-Feb;35(1):18-21, 29. PMID 26298938
- [Background] Vicariotto F. Effectiveness of an association of a cranberry dry extract, D-mannose, and the two microorganisms Lactobacillus plantarum LP01 and Lactobacillus paracasei LPC09 in women affected by cystitis: a pilot study. J Clin Gastroenterol. 2014 Nov-Dec;48 Suppl 1:S96-101. doi: 10.1097/MCG.0000000000000224. PMID 25291140
- [Background] Grin PM, Kowalewska PM, Alhazzan W, Fox-Robichaud AE. Lactobacillus for preventing recurrent urinary tract infections in women: meta-analysis. Can J Urol. 2013 Feb;20(1):6607-14. PMID 23433130